CLINICAL TRIAL: NCT05853692
Title: Prevention of Oral Mucositis in Subjects Undergoing Radiotherapy for Head and Neck Cancer. A Randomized Clinical Trial.
Brief Title: Prevention of Oral Mucositis in Head and Neck Cancer.
Acronym: OMHNC-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Prof., Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 4576
Record Dates: First submitted 2023-04-07; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a single-blind randomized clinical trial (RCT). The population will be divided into two groups, receiving respectively the medical device and a solution based on Sodium Bicarbonate (5 g/L)
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will be encharged of generating the allocation sequence, of enrolling the participants and of assigning the interventions to the participants.
  The coworkers who will evaluate the onset of OM and its severity will be blinded about the selected product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): The investigational product be administered for 63 days. Patient will use a spray based on zinc gluconate (three times a day)
  Interventions: Device: Zinc Gluconate
- Control (Active Comparator): The investigational product be administered for 63 days. Patient will use a solution based on sodium chloride and bicarbonate (5 times a day)
  Interventions: Device: Sodium Bicarbonate

INTERVENTIONS:
Device: Zinc Gluconate — Three times a day (spray)
  Arms: Test
Device: Sodium Bicarbonate — Five times a day (rinse)
  Arms: Control

SUMMARY:
Oral Mucositis (OM) consists in the painful inflammation and ulceration of the mucous membranes lining the digestive tract, lasting between 7 and 98 days; and starts as an acute inflammation of oral mucosa, tongue, and pharynx after RT exposure.

Gel X spray is a product based on zinc gluconate. It could be helpful to achieve the prevention of Oral Mucositis and, in case of OM manifestation, the reduction of oral pain symptoms and to accelerate the healing process of oral mucositis ulcerations.

The aim of this study is to demonstrate the efficacy of the treatment with Gel X to reduce the incidence of oral mucositis, in comparison with Sodium Bicarbonate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of the following HNC: oral cavity, pharynx, unknown primary, salivary glands, undergoing local radiotherapy for curative purpose
* Patients with diagnosis of HNC: oral cavity, pharynx, unknown primary, salivary glands, undergoing local radiotherapy as an adjuvant to surgical resection
* Patients able self-apply the product.

Exclusion Criteria:

* Patients with documented contraindication to any of the components of "Gel X" (there included eccipients): water, saccharin sodium, PVP, Taurine, Zinc Gluconate, PEG-40, Hydrogenated castor oil, Pullulan, Flavors
* Patients with any neurological and psychiatric condition having an influence on the ability to self-apply the treatment
* Patients participating to other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis | One week after the end of Radiotherapy
  Yes/No

SECONDARY OUTCOMES:
Time of Oral Mucositis Onset | From Day 0 to 2 months
  Days
Severity of Oral Mucositis | One week after the end of Radiotherapy
  Difference in Oral Mucositis Grade

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Hearth, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided